CLINICAL TRIAL: NCT01837602
Title: Clinical Trial of Autologous cMet Redirected T Cells Administered Intratumorally in Patients With Breast Cancer
Brief Title: cMet CAR RNA T Cells Targeting Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 13111, 813858
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2018-10

CONDITIONS: Metastatic Breast Cancer; Triple Negative Breast Cancer
Keywords: refractory to at least one standard therapy; newly diagnosed; with operable triple negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cMet positive breast cancer patients (Experimental): Metastatic breast cancer patients with an accessible tumor (cutaneous, subcutaneous, or superficial) and/or a palpable adenopathy/mass, with ≥ 30% tumor cells expressing cMet as demonstrated on immunohistochemical analysis . The intensity for cMet IHC should be greater than or equal to 1+. The targeted tumor must be accessible (i.e. is not near a great vessel or the spinal cord) and can be surgically excised or biopsied.
  Interventions: Biological: cMet RNA CAR T cells

INTERVENTIONS:
Biological: cMet RNA CAR T cells

SUMMARY:
An open-label, clinical trial of autologous cMet redirected T cells administered intratumorally (IT) in patients with breast cancer. Fifteen evaluable patients will be enrolled in stepwise fashion. Step 1 will enroll patients with metastatic breast cancer refractory to at least 1 standard therapy, step 2 will include newly diagnosed patients with operable triple negative breast cancer.

DETAILED DESCRIPTION:
This study is designed to determine the safety and feasibility of intratumoral administration of autologous T cells that have had genetic material transferred into the cell to redirect them to target breast cancer cells rather than their usual target. Eligible subjects will have metastatic breast cancer refractory to at least one standard therapy or to newly diagnosed with operable triple negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Step 1 subjects only: metastatic breast cancer patients with an accessible tumor (cutaneous, subcutaneous, or superficial) and/or palpable adenopathy/mass. The targeted tumor is accessible (i.e. is not near a great vessel or the spinal cord) and can be surgically excised or biopsied.
* Step 2 subjects only: Newly diagnosed, operable, triple negative breast cancer, i.e. ER/PR-negative, her2/neu-negative, with tumor size between 2 - 3 cm (T2) as measured by either clinical breast exam, mammogram, ultrasound or MRI, with or without ipsilateral axilla node involvement (N0 or N1).
* cMet expression in ≥ 30% tumor cells as demonstrated on immuno-histochemistry analysis of archival slides. The intensity for cMet IHC should be greater than or equal to 1+. Punch biopsy or percutaneous core biopsy may be offered to Cohort 1 patients. To establish eligibility for patients in step 1, archival tumor tissues from any previously biopsied metastatic tumor deposit may be used for IHC staining. The metastatic tumor nodule to be targeted for IT injection may not necessarily be the same as previously biopsied metastatic site.
* Age > 18 years old
* Baseline Eastern Cooperative Oncology Group (ECOG) Clinical Performance Status 0 or 1
* Adequate hematologic function:

WBC > 3.0 Plt > 75,000 Hgb > 10 g/dl Adequate renal function defined as serum creatinine < 1.5 times upper limit of normal

- Adequate hepatic function defined as: Total bilirubin < 1.5 times upper limit of normal, and ALT and AST < 2.5 times upper limit of normal

* Women of child bearing potential must have a negative pregnancy test (blood or urine) and agree to use appropriate contraception from study screen through the duration of the trial. Men must agree to use appropriate contraception from IT injection through the duration of the trial.
* Signed and dated written informed consent.

Exclusion Criteria:

* Step 1 subjects only: Targeted tumor near a great vessel or spinal cord
* Step 2 subjects only: Women already undergoing neoadjuvant chemotherapy to treat their primary triple negative breast cancer
* Step 1 and 2 subjects:Positive for HIV-1/HIV-2
* Active hepatitis B or hepatitis C infection
* The anticipated use of the following within 2 weeks prior to apheresis and prior to planned IT T-cell injection:

Immunosuppressive drugs Cytotoxic chemotherapy (See Section 5.7 for complete details) Systemic glucocorticoids (steroid prep due to dye allergies prior to staging scans or use in anti-emetic prophylaxis for patients undergoing chemotherapy is allowed) Hematopoietic growth factors Other experimental therapy Note: Step 1 patients receiving non-investigational targeted therapy (lapatinib, trastuzumab, and/or pertuzumab) are eligible provided these medicines are at a stable dose and the patient began taking them more than 30 days prior to the planned IT T-cell injection.

* Anticipated use of anti-coagulants such as coumadin, heparin, or Lovenox within 14 days before the planned IT T-cell injection RETIRED AS OF PROTOCOL VERSION 11
* Pregnant women or nursing mothers
* History of alcohol abuse or illicit drug use within 12 months of IT T-cell injection
* Clinically significant comorbid disease or other underlying condition, including major autoimmune disorders that would contraindicate study therapy or confuse interpretation of study results
* Significant psychiatric disorder and any other reason that in the Investigator's opinion would jeopardize protocol compliance or compromise the patient's ability to give informed consent.
* Prior MI ascertained from medical history and review of systems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-04; Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
Number of Serious Adverse Event | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Julia Tchou, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Tchou J, Zhao Y, Levine BL, Zhang PJ, Davis MM, Melenhorst JJ, Kulikovskaya I, Brennan AL, Liu X, Lacey SF, Posey AD Jr, Williams AD, So A, Conejo-Garcia JR, Plesa G, Young RM, McGettigan S, Campbell J, Pierce RH, Matro JM, DeMichele AM, Clark AS, Cooper LJ, Schuchter LM, Vonderheide RH, June CH. Safety and Efficacy of Intratumoral Injections of Chimeric Antigen Receptor (CAR) T Cells in Metastatic Breast Cancer. Cancer Immunol Res. 2017 Dec;5(12):1152-1161. doi: 10.1158/2326-6066.CIR-17-0189. Epub 2017 Nov 6. PMID 29109077